CLINICAL TRIAL: NCT02255370
Title: Controlled, Randomized, Double Blind Study, Comparing Curcumin to Thiopurines in the Prevention of Post-op Recurrence in Crohn Disease
Brief Title: Curcumin Associated With Thiopurin in the Prevention of Post-op Recurrence in Crohn Disease
Acronym: POPCUR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: 3i nature (Other); Naturopôle Nutrition santé (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0207; 2014-000261-51 (EudraCT Number)
Record Dates: First submitted 2014-09-19; First posted 2014-10-02 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Crohn's Disease
Keywords: Curcumin. Crohn's disease. Post-operative recurrence. Thiopurines . Rutgeerts endoscopic score
MeSH Terms: conditions — Crohn Disease | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- CURCUMIN (Experimental): subjects will be randomized into two arms; they will be given either placebo or curcumin 3g/d per os plus thiopurines during 6 months in a double-blind manner. Rutggerts endoscopic score at 6 months will be the main judgment criteria
  Interventions: Drug: Curcumin
- PLACEBO (Placebo Comparator): subjects will be randomized into two arms; they will be given either placebo or curcumin 3g/d per os plus thiopurines during 6 months in a double-blind manner. Rutggerts endoscopic score at 6 months will be the main judgment criteria
  Interventions: Drug: Curcumin

INTERVENTIONS:
Drug: Curcumin — subjects will be randomized into two arms; they will be given either placebo or curcumin 3g/d per os plus thiopurines during 6 months in a double-blind manner. Rutggerts endoscopic score at 6 months will be the main judgment criteria
  Other Names: placebo

SUMMARY:
Curcumin, the active ingredient of turmeric, has been used for long term in the treatment of inflammatory conditions. Inhibition of NF-κB is postulated as the main mechanism responsible for the anti-inflammatory effect of curcumin

Aim : to study the effect of curcumin, 3g per day, as compared to placebo, combined with thiopurines in the prevention of Crohn's disease post-operative recurrence.

DETAILED DESCRIPTION:
122 subjects, operated on for Crohn disease, will be included in the study. After ileo-colonic resection, subjects will be randomized into two arms; they will be given either placebo or curcumin 3g/d per os plus thiopurines during 6 months in a double-blind manner. Rutggerts endoscopic score at 6 months will be the main judgment criteria.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease confirmed by radiographic, endoscopic or histologic criteria
* Age > 18 yr
* Affiliated to french health insurance
* Operated on less than 15 days ago for ileal, colonic or ileo-colonic Crohn's disease with all macroscopic lesions being removed, with an anastomosis which can be reached by ileocolonoscopy

Exclusion Criteria:

* Ulcerative colitis
* Pregnant or nursing woman
* Refusal of contraceptive measure for childbearing potential, woman or fertile man
* Indication of anti-TNFα treatment
* Concomitant treatment including antibiotics, probiotics, mesalazine, methotrexate, cyclosporine, tacrolimus, anti-TNFα, ustekinumab, vedolizumab
* Concomitant treatment with corticosteroids, except in case of tapering a treatment initiated before surgery
* Renal insufficiency ( serum creatinine 2N)
* Chronic hepatic disease except for primary sclerosing cholangitis
* ALAT , ASAT, alkaline phosphatases, or bilirubin > 3N
* Current infection to HIV, HBV (except if HBV Ac positives), HCV
* Contraindication to thiopurines
* Unwillingness of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Rutgeerts endoscopic score | at 6 months

SECONDARY OUTCOMES:
CDAI score | at 6 months and at 1 year
Rutgeerts endoscopic score according to smoking status (yes/no) | at 6 months
Rutgeerts endoscopic score according to previous intestinal surgery (yes/no) | at 6 months
Rutgeerts endoscopic score according to anoperineal lesions (yes/no) | at 6 months
Rutgeerts endoscopic score according to a fistulising phenotype (yes/no) | at 6 months
Rutgeerts endoscopic score according to length of intestinal resection >0.5m | at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France